CLINICAL TRIAL: NCT06075745
Title: Cytomegalovirus (CMV) Vaccine in Orthotopic Liver Transplant Candidates (CTOT-44)
Brief Title: Cytomegalovirus (CMV) Vaccine in Orthotopic Liver Transplant Candidates
Acronym: COLT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT CTOT-44
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant
Keywords: Cytomegalovirus; Vaccine; Orthotopic Liver Transplant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccine Arm (Experimental): Participants in this arm will receive two doses of Cytomegalovirus-Modified Vaccinia Ankara (CMV-MVA) Triplex CMV vaccine
  Interventions: Drug: CMV-MVA Triplex
- Placebo Arm (Placebo Comparator): Participants will receive two doses of matching placebo of the Cytomegalovirus-Modified Vaccinia Ankara (CMV-MVA) Triplex CMV vaccine
  Interventions: Drug: Placebo for CMV-MVA Triplex

INTERVENTIONS:
Drug: CMV-MVA Triplex — The dosage used will be 5.0 x 10^8 pfu, administered under sterile conditions intramuscularly. The CMV-MVA Triplex vaccine lots range in titre from 5.0 to 9.0 x 10^8 pfu/mL in a supplied volume of 1.0 mL
  Arms: Vaccine Arm
Drug: Placebo for CMV-MVA Triplex — Arm 2 participants receive two doses of matching placebo CMV-MVA Triplex
  Arms: Placebo Arm

SUMMARY:
This is a multi-center clinical trial in Cytomegalovirus (CMV) seronegative prospective liver transplant recipients to determine the efficacy of two doses of Cytomegalovirus-Modified Vaccinia Ankara (CMV-MVA) Triplex CMV vaccine pre-transplant. The primary objective is to assess the effect of pre-transplant (Tx) Triplex vaccination on duration of CMV antiviral therapy (AVT) within the first 100 days post-Tx in CMV seropositive donor (D+) and seronegative (R-) (D+R-) liver transplant recipients (LTxRs). A protocol-mandated preemptive therapy (PET) will be used for CMV disease prevention in D+R- LTxRs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and provide informed consent
2. Negative for Cytomegalovirus (CMV) IgG antibody as assessed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory within 12 months of enrollment, and no history of prior positive CMV serology (IgG antibody)
3. Negative human immunodeficiency virus (HIV) testing and no clinical suspicion of HIV infection
4. Planned for a first living donor liver transplant or listed/anticipated to be listed for a first deceased donor liver transplant.
5. Anticipated to receive a liver transplant within 1-12 months
6. For individuals of reproductive potential, a negative serum or urine pregnancy test within 72 hours prior to enrollment. NOTE: Individuals of reproductive potential are defined as individuals who have reached menarche and who have not been post-menopausal for at least 12 consecutive months with follicle-stimulating hormone (FSH) >=40 IU/mL or 24 consecutive months if an FSH is not available, i.e., who have had menses within the preceding 24 months, and have not undergone a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, or salpingectomy)
7. Participants who are able to impregnate or become pregnant (i.e., of reproductive potential) and are participating in sexual activity that could lead to pregnancy must agree to practice contraception/birth control (hormonal or barrier method) or agree to not participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) for at least 1 month following the last vaccine/placebo dose. For acceptable contraception methods that are more than 80 percent effective, see Food and Drug Administration (FDA) Office of Women's Health (http://www.fda.gov/birthcontrol)
8. The most recent platelet count is >= 20,000 cells/mm^3 within 3 months prior to enrollment and in the opinion of the investigator, has not decreased < 20,000 cells/mm^3 at time of study IP administration.

Eligibility criteria required: Dose 2:

1. Most recent platelet count >= 20,000 cells/mm^3 within 3 months prior to enrollment and in the opinion of the investigator, has not decreased < 20,000 cells/mm^3 since last result
2. For women of reproductive potential as defined previously, a negative serum or urine pregnancy test (performed within 72 hours)

Exclusion Criteria:

1. Women who are breastfeeding or planning to breastfeed
2. Prior Cytomegalovirus (CMV) vaccination
3. Receipt of immunoglobulin or CMV-specific immunoglobulin within the last 3 months (this includes coronavirus disease (COVID) convalescent plasma)
4. Currently enrolled in another interventional study that, in the investigator's opinion, could affect the evaluation of safety and/or vaccine effect outcomes
5. Prior (ever) receipt of a stem cell transplant (Peripheral blood stem cell (PBSC), marrow, cord blood, etc.)
6. Receipt of immunosuppression:

   * Within the last 3 months prior to randomization:

     * Systemic Chemotherapy or immunotherapy for cancer in the last 3 months (localized therapy for hepatocellular carcinoma [HCC] such as chemoembolization, Y-90 are not considered "systemic chemotherapy" and are not excluded)
     * Systemic immunosuppressive agents (e.g., cyclophosphamide, methotrexate, mycophenolate, azathioprine, calcineurin inhibitors, mTOR inhibitors, TNF-alpha inhibitors) and/or combination immunosuppressive drugs for any autoimmune or other conditions in the last 3 months except corticosteroids as below
   * Within the last 28 days prior to randomization: averaged daily corticosteroid therapy dose ≥20 mg of prednisone equivalent
   * Within the last 6 months prior to randomization: receipt of T- or Bcell depleting agents (e.g. ATG, Alemtuzumab, Rituximab)
7. Transplant status 1A or in the opinion of the investigator is likely to receive a transplant within the next month
8. At the time of randomization, either listed for, or, in the opinion of the investigator, likely to receive any non-liver organ transplant
9. Receipt of a clinical vaccine < 14 days before or planned to receive a clinical vaccine <14 days after the study agent
10. Known allergy to any component of the study agent
11. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Exclusion criteria required: Dose 2:

1. Anaphylaxis or other severe reaction (Grade 4) considered definitely or probably attributable to dose 1
2. Receipt of liver transplant prior to dose 2
3. The participant must not have any severe acute illness or other factor, that, in the opinion of the investigator, requires postponement of dose 2 because of safety concerns. The participant can be re-evaluated for eligibility throughout the window of eligibility for the dose 2, once the illness or other factor has improved or resolved
4. Receipt of a clinical vaccine < 14 days before or planned to receive a clinical vaccine <14 days after the study agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Total days of Cytomegalovirus (CMV) active antiviral therapy (AVT) in CMV seropositive donor (D+) and seronegative (R-) and (D+R-) liver transplant recipients | Within the first 100 days post-transplantation
Percent of participants with solicited adverse reactions | Within 7 days of each dose
  Consisting of local reactions including: injection site pain, swelling, erythema (redness); systemic reactions: fever, headache, muscle ache, fatigue)
Percent of participants with pre-transplant treatment emergent serious adverse events (TESAE) | Within 100 days after initial dose
Percent of participants with pre-transplant treatment emergent serious adverse events (TESAE) | Within 28 days after each dose
Percent of participants with pre-transplant treatment emergent adverse events (TEAE) | Within 28 days after each dose
  Grade >=3 severity or increase of severity of baseline abnormality that results in grade >= 3 severity
Percent of participants with treatment emergent serious adverse events (TESAE) | Throughout the study
  Grade >= 4 severity

SECONDARY OUTCOMES:
Percent of seropositive donor (D+) and seronegative (R-) liver transplant recipients (D+R- LTxRs) who develop Endpoint-Committee adjudicated Cytomegalovirus (CMV) disease | By 6 months post-transplant (Tx)
Percent of seropositive donor (D+) and seronegative (R-) liver transplant recipients (D+R- LTxRs) who develop investigator-reported Cytomegalovirus (CMV) disease | By 6 months post-transplant (Tx)
Time to onset of Endpoint-Committee adjudicated Cytomegalovirus (CMV) disease in seropositive donor (D+) and seronegative (R-) (D+R-) liver transplant recipients | By 6 months post-transplant (Tx)
Time to onset of Endpoint-Committee adjudicated Cytomegalovirus (CMV) in seropositive donor (D+) and seronegative (R-) (D+R-) liver transplant recipients | By 6 months post-transplant (Tx)
Time to onset of investigator-reported Cytomegalovirus (CMV) disease | By 6 months post-transplant (Tx)
Percent of seropositive donor (D+) and seronegative (R-) liver transplant recipients (D+R- LTxRs) who develop CMV DNAemia >= 1000 IU/mL | Within first 100 days post-transplant (Tx)
Percent of seropositive donor (D+) and seronegative (R-) liver transplant recipients (D+R- LTxRs) who develop Endpoint committee adjudicated CMV disease | Within first 100 days post-transplant (Tx)

CONTACTS AND LOCATIONS:
Overall Officials: Ajit P Limaye, MD, Study Chair — University of California, San Francisco: Transplantation; Cindy Fisher, M.D., Study Chair — University of Washington Medical Center: Transplantation
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, School of Medicine, Birmingham, Alabama
  - University of California, San Diego School of Medicine, La Jolla, California
  - Stanford University, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester - College of Medicine and Science, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University School of Medicine, Durham, North Carolina
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Medical Center: Transplantation, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial
Access Criteria: Open access
URL: http://www.immport.org/home

REFERENCES:
- See also: Clinical Trials in Organ Transplantation — http://www.ctotstudies.org
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait